CLINICAL TRIAL: NCT06168630
Title: Effects of Manual Lymph Drainage on Breast Engorgement, Pain and Self Efficacy in Postpartum Period.
Brief Title: Effects of Manual Lymph Drainage on Breast Engorgement in Postpartum Period.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Adeela Arif, Senior Lecturer, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aqsa Ejaz
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Postpartum
Keywords: Engorgement; Manual lymph drainage; Postpartum period; Pain; Self efficacy
MeSH Terms: conditions — Hyperemia; Pain | interventions — Manual Lymphatic Drainage; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymph Drainage (Experimental)
  Interventions: Other: Manual lymph drainage
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Manual lymph drainage — It consists of patients who will receive manual lymph drainage everyday for 5 days. The subject's position will be supine with their knees bent. Every session will be of 45 minutes. Manual lymph drainage will with abdominal lymph drainage, after which central lymph stimulation will be performed. Then, by stimulating the bilateral axillary lymph nodes, the flow of fluid over the right and left breasts will be directed toward the axillary lymph nodes. While the patients in the prone position, bilateral axillary lymph nodes will be stimulated, and each manual lymph drainage will be performed from the dorsum to the axillary lymph node .
  Arms: Manual Lymph Drainage
Other: Control group — The other group will receive massage for 20 minutes every day for 5 days from first day of treatment. Massage will be done using the index and middle fingers in a spiral motion towards the nipples.
  Arms: Control group

SUMMARY:
There have been many studies on the treatment of breast engorgement, there is a lack of research comparing the effectiveness of manual lymph drainage with massage. Therefore, this study will be a randomized controlled trial that aims to compare the effects of manual lymph drainage with massage on breast engorgement, pain, and self efficacy in the postpartum period.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial and will be conducted in Jinnah hospital, Lahore. This study will be completed in time duration of 10 months after the approval of synopsis. Non probability convenience sampling technique will be used and 35 participants will be recruited in study after randomization. The subjects will be divided into two groups and the group A will receive manual lymph drainage and group B will receive massage whereas cold pack will be used as a baseline treatment. The tools that will be used for pre and post treatment assessment are NPRS, 6 point self rated engorgement scale and breast feeding self efficacy questionnaire. The data will be assessed after 5 days of treatment using 2 tailed t test. After data collection data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

Women aged 25 to 35 years. Lactating mothers who presents with breast pain after birth. Women with breast heaviness. Women who rate themselves 4 on engorgement scale on six-point self-rated engorgement scale.

Exclusion Criteria:

Patients with gastrointestinal, urogynaecological, autoimmune or any neurological condition.

Women with breast cancer. Women with breast abcess. Women taking other medications.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | 5th day
  The Numerical pain rating scale is the most commonly used pain scale in the health care.
  This scale is used on subjects of age more than 9. By using this scale ask the participant to rate their pain orally by giving the numbers from 0-10
Six point self rated engorgement scale | 5th day
  Six point self rated engorgemet scale is valid and reliable measures to assess breast engorgement and pain
Breast feeding self efficacy questionnaire | 5th day
  The divergent validity of the BSES-SF was proved via a significant negative correlation with scores of the Edinburgh Postnatal Depression Scale (r = - 0.273, P < 0.001). BSES-SF is a reliable and valid instrument for measuring breastfeeding self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International university, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monazzami M, Yousefzadeh S, Rakhshandeh H, Esmaeili H, Afiat M. The effect of hot ginger compress (Zingiber officinale) on the severity of breast engorgement in lactating women. The Iranian Journal of Obstetrics, Gynecology and Infertility. 2019;21(12):77-84.
- [Background] Song JA, Hur MH. A Systematic Review of Breast Care for Postpartum Mothers. Korean J Women Health Nurs. 2019 Sep;25(3):258-272. doi: 10.4069/kjwhn.2019.25.3.258. Epub 2019 Sep 2. PMID 37679918
- [Background] Manna M, Podder L, Devi S. Effectiveness of hot fomentation versus cold compression on breast engorgement among postnatal mothers. International Journal of Nursing Research and Practice. 2016;3(1):13-8.